CLINICAL TRIAL: NCT03185923
Title: A Randomized Controlled Trial of Integrated Traditional Chinese and Western Medicine in the Treatment of Severe Community Acquired Pneumonia
Brief Title: Effect of Traditional Chinese Medicine on Outcomes in Patients With Severe Pneumonia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for severe pneumonia
Record Dates: First submitted 2017-06-04; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Community-Acquired Infections
Keywords: Community-Acquired Infections; Humans; Medicine, Chinese Traditional
MeSH Terms: conditions — Community-Acquired Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM plus conventional drug (Experimental): The experimental group will receive three type of TCM inaddition conventional drug according to china CAP guidline 2016.
  Interventions: Drug: TCM plus conventional drug
- TCM placebo plus conventional drug (Placebo Comparator): The control group will receive three type of placebo TCM inaddition conventional drug according to china CAP guidline 2016.
  Interventions: Drug: TCM placebo plus conventional drug

INTERVENTIONS:
Drug: TCM plus conventional drug — All patients were treated with antibiotics according to international guidelines. The Experimental group will receive TCM according to the TCM syndrome.
  qingfeijieduhuatan granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for phlegm-heat obstructing in the lung syndrome in 28 treatment days.
  zaoshihuatanxiefei granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for pulmonary stagnation of phlegm syndrome in 28 treatment days.
  qingxinkaiqiao granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for Pathogenic heat trapping the pericardium syndrome in 28 treatment days.
  shenmai injection（Sichuan chuanda west China Pharmaceutical Co., Ltd.）,15ml/ ampulla, 10～60ml each time (when needed), for yin exhausted syndrome in 28 treatment days.
  shenfu injection（Sanjiu Medical & Pharmaceutical Co., Ltd.）,10ml/ ampulla, 50～100ml each time (when needed), for yang exhausted syndrome in 28 treatment days.
  Arms: TCM plus conventional drug
Drug: TCM placebo plus conventional drug — All patients were treated with antibiotics according to international guidelines. The control group will receive TCM placebo according to the TCM syndrome.
  placebo qingfeijieduhuatan granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for phlegm-heat obstructing in the lung syndrome every day in 28 treatment days.
  placebo zaoshihuatanxiefei granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for pulmonary stagnation of phlegm syndrome every day in 28 treatment days.
  placebo qingxinkaiqiao granule (Sanjiu Medical & Pharmaceutical Co., Ltd.), 10g/packet, twice daily, for Pathogenic heat trapping the pericardium syndrome every day in 28 treatment days.
  Arms: TCM placebo plus conventional drug

SUMMARY:
This study evaluates the integrated traditional Chinese and Western medicine in the treatment of severe community acquired pneumonia in adults. Half of participants will receive traditional Chinese and Western medicine in combination, while the other half will receive a placebo traditional Chinese and Western medicine.

DETAILED DESCRIPTION:
Improving the care of patients with community-acquired pneumonia (CAP) has been the focus of many different organizations. Such efforts at improvement in care are warranted, because CAP, especially severe CAP remains the leading cause of death in the world. Despite advances in antimicrobial therapy, rates of mortality due to severe CAP have not decreased significantly since penicillin became routinely available.

traditional Chinese Medicine, has been used for thousands of years in treating pneumonia. To date, it has become popular and widely practiced in many countries around the world. In the past decades, Evidences from both clinicians and patients suggest that there is some beneficial effect of TCM on severe CAP.

At present, there are many therapies available for patients with severe CAP, it is difficult for us to identify the most suitable therapy. Thus, this study aims to compare the efficacy of combination conventional drug and TCM to the conventional drug and placebo, and then determine which one is the better therapy, providing a scientific basis for clinical decision.

This is a multi-center, randomized, controlled trial to compare the efficacy of two therapies for patients with severe CAP. 198 subjects will be randomly assigned to one therapies (conventional drug, and the combination of conventional drug and TCM) for 28 days treatment. After the treatment period, subjects in two arms will be followed up for 12 weeks. The primary outcomes will include treatment failure, and secondary outcomes Time to clinical stability, length hospital stays, in-hospital mortality, SOFA questionnaire, quality of life (CAP-PRO ) and health economics.

ELIGIBILITY:
Inclusion Criteria:

* were aged 18 years to 80 years.
* met severe community-acquired pneumonia criteria (defined by modified American Thoracic Society criteria).
* Syndrome differentiation meets criteria of phlegm-heat obstructing in the lung syndrome, pulmonary stagnation of phlegm syndrome, Pathogenic heat trapping the pericardium syndrome, or Pathogenic depression is taking off syndrome.

Exclusion Criteria:

* Pregnant and lactating women.
* trauma, hematologic malignancies, various solid tumors, and obstetric complications.
* Aspiration pneumonia, fungal pneumonia, HIV related Pneumocystis carinii pneumonia, tuberculosis, Bronchiectasis with infection and pulmonary abscess;
* Dementia, mental disorders and reluctant partners.
* Be discharged from hospital within 2 days or require operation.
* reported severe immunosupression (human immunodeficiency virus infection, immunosuppressive conditions or medications).
* Neuromuscular disorders affecting respiratory motor function.
* Patients with severe cardiovascular，with severe liver and kidney disease.
* Patients who have participated in other clinical studies in the past 4 weeks.
* Patients unwilling to sign informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-06-20 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | up to 28 days.
  The primary efficacy outcome was the rate of treatment failure, which includes treatment failure that occurred.

SECONDARY OUTCOMES:
time to clinical stability | up to 28 days.
  Clinical stability
length hospital stays | up to 28 days.
  length hospital stays will be recorded.
in-hospital mortality | up to 28 days.
  in-hospital mortality will be recorded.
SOFA questionnaire | Change from baseline SOFA score at day 0、7、14、28 of the treatment phase.
  Clinical symptom assessment questionnaire of severe CAP
CAP -CRO | Change from baseline CAP -CRO score at day 0、7、14、28 of the treatment phase.at week 4, week 8, week 12 of the follow-up phase.
  CAP doctor reported outcome scale will be used to assess symptoms.
Health economics | up to 28 days.
  Cost of the treatment phase will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Li J, Yu X, Li SY. Integrated traditional Chinese and conventional medicine in treatment of severe community-acquired pneumonia: study protocol for a randomized placebo-controlled trial. Trials. 2018 Nov 12;19(1):620. doi: 10.1186/s13063-018-3005-9. PMID 30419961